CLINICAL TRIAL: NCT06474182
Title: Comparison of the Effects of Prophylactic Administration of Apixaban on Thrombin Generation in Patients With de Novo Multiple Myeloma and Patients Undergoing a Surgery for Total Knee Replacement
Brief Title: Comparison of the Effects of Apixaban on Thrombin Generation in Patients With de Novo Multiple Myeloma
Acronym: ProApix
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23CH293; ANSM (Other: 2024-A00769-38)
Record Dates: First submitted 2024-04-23; First posted 2024-06-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Total Knee Replacement
Keywords: Multiple myeloma; thromboprophylaxis; pharmacodynamics; coagulability
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection; apixaban

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood sampling of patients with de novo multiple myeloma (Experimental): Description: Blood sampling of patients with de novo multiple myeloma
  Interventions: Procedure: Blood sampling; Drug: Apixaban
- Blood sampling of patients undergoing total knee replacement (Experimental): Description: Blood sampling of patients undergoing total knee replacement
  Interventions: Procedure: Blood sampling; Drug: Apixaban

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling
Drug: Apixaban — Treatment by Apixaban

SUMMARY:
Patients with multiple myeloma (MM) are at high risk of venous thromboembolism (VTE) and these patients require adequate thromboprophylaxis. Following the publication of the AVERT clinical study, Apixaban is strongly recommended as a prophylactic treatment option for patients with cancer, based on high quality of evidence and a favorable efficacy/safety profile. A multicenter and ancillary study - APIXABOR - that measured the plasmatic concentration of Apixaban in patients with MM and treated with preventive dose has been conducted. The peak drug concentration was superior in MM plasma, as compared to non-myeloma patients under prophylaxis. Therefore, the present study evaluated whether differences in pharmacokinetics have an impact on pharmacodynamics (i.e. decrease in coagulability in MM patients as compared to non-MM patients undergoing a surgery for total knee replacement who also have VTE prophylaxis). In fine, this study may inform to better manage thromboprophylaxis in MM patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Signed informed consent,
* Patient covered by a social security scheme.
* Group 1 : patient with a diagnosis of de novo multiple myeloma, with an indication of thromboprophylaxis with Apixaban,
* Group 2 : patient requiring a surgery for total knee replacement, , with an indication of thromboprophylaxis with Apixaban.

Exclusion Criteria:

* Curative doses of anticoagulation treatment,
* Contra-indication to Apixaban,
* Pregnant or breastfeeding woman,
* Refusal to sign consent,
* Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Endogenous Thrombin potential (nM.min) | 2 hours after Apixaban Treatment
  Endogenous Thrombin potential (nM.min) as measured with MidiCAT method at the concentration peak 2 hours after 2.5mg Apixaban treatment

SECONDARY OUTCOMES:
Apixaban concentration (ng/mL) | Kinetics of 12 hours following Apixaban treatment in both groups
  Apixaban concentration (ng/mL) as measured by mass spectrometry during 12 hours following Apixaban treatment (2.5mg) in both groups
Pharmacodynamics' kinetics of Endogenous Thrombin Potential | Kinetics of 12 hours following Apixaban treatment in both groups
  MidiCAT method measure : Endogenous Thrombin Potential (nM.min)
Pharmacodynamics' kinetics of Lagtime | Kinetics of 12 hours following Apixaban treatment in both groups
  MidiCAT method measure : Lagtime (min)
Pharmacodynamics' kinetics of Time to peak | Kinetics of 12 hours following Apixaban treatment in both groups
  MidiCAT method measure : Time to peak (min)
Pharmacodynamics' kinetics of Thrombin peak | Kinetics of 12 hours following Apixaban treatment in both groups
  MidiCAT method measure : Thrombin peak (M, Thrombin)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CHALAYER, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France